CLINICAL TRIAL: NCT01706588
Title: Preliminary Evaluation of the Efficacy and Local Tolerability of Injectable Diclofenac at 5, 12.5, 25 and 50 mg/mL, Administered Locally Prior to Surgery for the Prevention of Post-operative Pain After Third Molar Surgery
Brief Title: Injectable Diclofenac for the Prevention of Post-operative Dental Pain
Acronym: DP4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12UK/DCsc04
Record Dates: First submitted 2012-10-01; First posted 2012-10-15 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Pain
Keywords: diclofenac, postsurgical pain, oral surgery
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Diclofenac sodium 5 mg/mL (Experimental)
  Interventions: Drug: Diclofenac sodium
- Diclofenac sodium 12.5 mg/mL (Experimental)
  Interventions: Drug: Diclofenac sodium
- Diclofenac sodium 25 mg/mL (Experimental)
  Interventions: Drug: Diclofenac sodium
- Diclofenac sodium 50 mg/mL (Experimental)
  Interventions: Drug: Diclofenac sodium
- Placebo 1 mL (Placebo Comparator)
  Interventions: Drug: Diclofenac sodium

INTERVENTIONS:
Drug: Diclofenac sodium — One single diclofenac injection into the surgical area before surgery but as soon as the anaesthetic has taken effect.
  Other Names: Diclofenac HPBCD

SUMMARY:
This is a prospective, randomised, double-blind, placebo-controlled, parallel group study in approximately 75 patients undergoing surgical removal of an impacted lower third molar.

ELIGIBILITY:
Inclusion Criteria:

1. Out-patients of either gender.
2. Patients aged ≥ 18 to ≤ 65 years old.
3. Subjects able and willing to give their written consent prior to inclusion in the study.
4. Female subjects of childbearing potential must (1) have a negative urine pregnancy test at the inclusion visit, (2) be using an appropriate method of contraception according to the definition of Note of ICH M3 Guideline (implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner), and (3) be willing to continue using the contraceptive method throughout the entire study period.
5. Subjects must (1) be able to comprehend the full nature and purpose of the study, including possible risks and side effects, (2) fully co-operate with the Investigator, (3) comply with the requirements of the entire study.
6. Patients undergoing surgical extraction of a single, fully or partially impacted mandibular 3rd molar requiring bone removal.

Exclusion Criteria:

General

1. Patients refusing to give written informed consent.
2. Patients not able to understand the purposes of the study or not willing to return for the control visits.
3. Patients with major psychiatric disorders that, in the investigator's opinion, could compromise study participation.
4. Patients enrolled in any clinical trial in the previous 3 months.
5. Employees of the study centre with direct involvement in the proposed study or other studies under the direction of the main investigator or study centre, as well as family members of the employees or investigator.
6. Pregnant or breast-feeding women.
7. Alcohol or drug abuse in the previous 12 months.
8. Clinically significant or unstable concomitant disease whose sequelae might interfere with the study evaluation parameters.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dietrich, MD, Principal Investigator — The School of Dentistry, University of Birmingham
Locations (1):
- The School of Dentistry University of Birmingham, Birmingham, United Kingdom

REFERENCES:
- [Derived] Gorecki P, Rainsford KD, Taneja P, Bulsara Y, Pearson D, Saund D, Ahmed B, Dietrich T. Submucosal Diclofenac for Acute Postoperative Pain in Third Molar Surgery: A Randomized, Controlled Clinical Trial. J Dent Res. 2018 Apr;97(4):381-387. doi: 10.1177/0022034517744207. Epub 2017 Dec 4. PMID 29202646

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo 1 mL: One single placebo injection into the surgical area before surgery but as soon as the anaesthetic has taken effect.
Period: Overall Study
Arm/Group | Diclofenac Sodium 5 mg/mL | Diclofenac Sodium 12.5 mg/mL | Diclofenac Sodium 25 mg/mL | Diclofenac Sodium 50 mg/mL | Placebo 1 mL
Started | 15 | 15 | 15 | 14 | 16
Completed | 15 | 15 | 15 | 14 | 16
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Sodium 5 mg/mL | Diclofenac Sodium 12.5 mg/mL | Diclofenac Sodium 25 mg/mL | Diclofenac Sodium 50 mg/mL | Placebo 1 mL | Total
Number analyzed (Participants) | 15 | 15 | 15 | 14 | 16 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7.3) | 28 (9.4) | 30 (9) | 27 (4.5) | 30 (9.5) | 28.6 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 12 | 8 | 12 | 47
  Male | 6 | 9 | 3 | 6 | 4 | 28

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of the Pain Scores.
Description: Pain will be scored by the patient at the end of surgery (time 0) and at 15-minute intervals after surgery for a total of 6 hours on a 0-100 mm VAS (from 0 = no pain to 100 = worst pain imaginable).
Time Frame: Pain scores will be measured over the time from end of surgery (time 0) to the 6 hour post-surgery
Measure: Mean (Standard Deviation); unit: mm*minutes
Arm/Group | Diclofenac Sodium 5 mg/mL | Diclofenac Sodium 12.5 mg/mL | Diclofenac Sodium 25 mg/mL | Diclofenac Sodium 50 mg/mL | Placebo 1 mL
Number analyzed (Participants) | 15 | 15 | 15 | 14 | 16
mm*minutes | 6843 (6259) | 8832 (6330) | 9998 (8080) | 7290 (6509) | 15539 (9279)

2. Secondary Outcome: Postsurgical Extra-oral Swelling
Time Frame: measured at 6 hours postsurgery, at day 3 and 1 week postsurgery
Reporting Status: Not Posted

3. Secondary Outcome: Trismus
Time Frame: measured at 6 hours postsurgery, at day 3 and 1 week postsurgery
Reporting Status: Not Posted

4. Secondary Outcome: Peak Pain Intensity
Time Frame: measured from end of surgery up to 12 hours postsurgery
Reporting Status: Not Posted

5. Secondary Outcome: Time to First Use of Rescue Medication.
Time Frame: measured from end of surgery up to 1 week postsurgery
Reporting Status: Not Posted

6. Secondary Outcome: Amount of Rescue Medication
Time Frame: consumed by the patient every 15-minutes postsurgery up to 6 hours postsurgery
Reporting Status: Not Posted

7. Secondary Outcome: Rescue Medication Consumption
Time Frame: consumed by the patient from end of surgery up to 24 and up to 48 hours postsurgery
Reporting Status: Not Posted

8. Secondary Outcome: Patient and Investigator Global Evaluation of the Effectiveness of Treatment
Time Frame: at 6 hour postsurgery and on Day 3
Reporting Status: Not Posted

9. Secondary Outcome: Time to Onset of Pain
Time Frame: measured from end of surgery up to 12 hours postsurgery
Reporting Status: Not Posted

10. Secondary Outcome: Wound Healing
Time Frame: at 6 hour postsurgery, and on day 3 and 1 week postsurgery
Reporting Status: Not Posted

11. Secondary Outcome: Recurrent Bleeding
Time Frame: every hour up to 6 hour postsurgery
Reporting Status: Not Posted

12. Secondary Outcome: Vital Signs
Time Frame: presurgery (within 30 days from surgery), at day of surgery (day 1), day 3 and 1 week postsurgery.
Reporting Status: Not Posted

13. Secondary Outcome: Number of Patients With Adverse Events
Time Frame: from signature of the informed consent to 1 week postsurgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Diclofenac Sodium 5 mg/mL | Diclofenac Sodium 12.5 mg/mL | Diclofenac Sodium 25 mg/mL | Diclofenac Sodium 50 mg/mL | Placebo 1 mL
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 6/15 | 7/15 | 5/15 | 5/14 | 6/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium 5 mg/mL (N=15) | Diclofenac Sodium 12.5 mg/mL (N=15) | Diclofenac Sodium 25 mg/mL (N=15) | Diclofenac Sodium 50 mg/mL (N=14) | Placebo 1 mL (N=16)
ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
injection site pain (General disorders) | 2 (2) | 2 (2) | 4 (5) | 1 (1) | 0 (0)
swelling (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
injection site swelling (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
linphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
gingival ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less